CLINICAL TRIAL: NCT04635657
Title: Pre and Post-Operative Cognitive Status in Patients Undergoing Surgery for Resection of Meningioma Associated With the Frontal and Temporal Lobes
Brief Title: Cognitive Status After Removal of Skull Base Meningioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel M. Prevedello, Clinical Professor, Ohio State University
Other Study IDs: 2019H0340
Record Dates: First submitted 2020-09-29; First posted 2020-11-19 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Meningioma; Skull Base Meningioma; Frontal Meningioma; Temporal Meningioma; Cognitive Impairment; Cognitive Decline; Post-Surgical Cognition
MeSH Terms: conditions — Meningioma; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meningioma Group: This group will include all patients in the study, regardless of location (frontal or temporal lobe) or surgical approach (endoscopic endonasal or craniotomy). Fifty patients will be included in the cohort
  Interventions: Other: Long-term Cognitive testing

INTERVENTIONS:
Other: Long-term Cognitive testing — These patients will undergo their standard of care cognitive testing at baseline, six weeks post-operatively and one year post-operatively.

SUMMARY:
The purpose of this prospectively enrolling trial is to assess long-term cognitive outcomes of patients undergoing surgery for resection of a meningioma associated with the frontal and temporal lobes.

DETAILED DESCRIPTION:
This study will look at patients who are undergoing resection of a skull based meningioma, located in the frontal or temporal lobe, via craniotomy or via endoscopic endonasal approach. The study will compare cognitive function at baseline, at six weeks postoperatively and at one year postoperatively. The cognitive testing being done at baseline will be a clinical care set of assessments done by the speech language pathology team and will include the RBANS tests, the MoCA, PROMIS-29, and NeuroQOL-Cognitive Functions.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a meningioma associated with the frontal or temporal lobes
* Subject is scheduled to undergo open craniotomy or Endoscopic Endonasal surgery
* Subject is 18 years of age or older
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent
* Previous surgery will not exclude the patient as a new baseline cognitive evaluation will occur.

Exclusion Criteria:

* Patient is a prisoner
* Patient is 90 years of age or older
* Pregnant women
* Previous radiation to the brain

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between 18 years of age and 89 years of age will be eligible for this study. Patients undergoing a resection of a meningioma located in the frontal or temporal lobes via craniotomy or endoscopic endonasal surgery for clinical purposes will be included. Should a patient have a previous surgical removal of a meningioma, they will still be included. However, all patients having undergone previous radiation to the brain, for any reason, will not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall cognitive function | 12 months
  Cognitive function will be compared at baseline and at one year post-operatively.

SECONDARY OUTCOMES:
Cognitive function based on surgical approach using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12 months
  Patients divided by approach and overall cognitive function will be evaluated.
Cognitive function based on tumor location using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12 months
  Patients will be divided by tumor location and cognitive function will be evaluated.

OTHER OUTCOMES:
Surgical comorbidities based on quality of life questionnaire PROMIS-29 | 12 months
  Assessment of preoperative and postoperative comorbidities and their effects on cognitive function post-operatively. Co-morbidities will be based on clinical outcomes evaluated by the primary investigator, co-investigators and the speech language pathology team.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Prevedello, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There will not be sharing of individual participant data with other researchers